CLINICAL TRIAL: NCT04383769
Title: Differentiated Service Delivery for Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: DSD-ART
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 5,000 participants:: 2,500 are PLHIV receiving standard care in the hospital and 2,500 are PLHIV receiving care in DSD-ART model
  Inclusion criteria:
  1. Thai citizenship
  2. Age ≥ 18
  3. HIV positive
  4. Received ART for at least 6 months at a participating hospital (Except for After hour ART clinic model that will allow participants who receive ART less than 6 months into service)
  5. One of the following:
     1. Accept DSD-ART, OR
     2. Already receiving DSD-ART, OR
     3. Decline DSD-ART and will continue standard ART service at the hospital.
  Interventions: Other: questionnaires survey

INTERVENTIONS:
Other: questionnaires survey — data will be collected from the medical records already existed in the hospital and community-based organization (CBO) systems and entered into case report form (CRF). The expected number of participants is 5000. For each participant, the data will be collected prospectively for 24 months and retrospectively up to 5 years from the screening date. This study has no intervention and will not alter ART services whether be standard or DSD-ART at hospitals.

SUMMARY:
This study is a prospective observational cohort. The target study population is PLHIV who receive ART at hospitals and community-based organizations (CBOs) in Chiang Mai, Ubon Ratchathani, Chonburi, and Songkhla. Participants will receive ART service in the same standard as in the hospital setting. Secondary data will be collected from the medical records already existed in the hospital and CBO systems.

DETAILED DESCRIPTION:
DSD-ART service at the Hospital

* Medical examination: All clients who receive ART service at the hospital and agree to participate in the research project will be interviewed to collect personal information and receive physical and laboratory examination in order to assess eligibility in research participation. If ineligible, the clients will be referred to the standard of care.
* Preparation and DSD-ART service offer: PLHIV who are eligible to participate in the research will receive counselling to assess the supports the clients need and will be offered various models of DSD-ART service. The clients may choose the model that is most suitable to their lifestyle.

ELIGIBILITY:
Inclusion Criteria:

1. Thai citizenship
2. Age ≥ 18
3. HIV positive
4. Received ART for at least 6 months at a participating hospital (Except for After hour ART clinic model that will allow participants who receive ART less than 6 months into service)

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data officer will collect secondary data regarding ART refill, laboratory test, counseling, doctor visit for HIV-related conditions, such as adverse drug reaction, opportunistic infections, and comorbidities, from the medical records already existed in the hospital and community-based organization systems and entered into the case report form. The identity of the clients will be untraceable since UL, which is a unique letter code assigned to each participant using Thai initials and date of birth translated into English alphabets, will be used as an individual identifier. The data will be collected prospectively for 24 months and retrospectively for up to 5 years from the screening date.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
differentiated service delivery for antiretroviral therapy (DSD-ART) | 5 years
  1. To assess retention among people living with HIV (PLHIV) in various models of differentiated service delivery for antiretroviral therapy (DSD-ART) Hypothesis: The proportions of PLHIV with high ART retention in each DSD-ART model are similar and not inferior to standard-of-care historical data

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD,Ph.D, Principal Investigator — Institute of HIV Research and Innovation (IHRI)
Locations (1):
- 3. Swing Dic,, Chon Buri, Thailand